CLINICAL TRIAL: NCT06608381
Title: Comparison Between Partial Omentectomy and Total Omentectomy During Minimally Invasive Radical Distal Gastrectomy for Clinical T3 and T4a Gastric Cancer; Multicenter Randomized Clinical Trial (KLASS-10)
Brief Title: Comparison Partial Versus Total Omentectomy in Minimal Invasive Distal Gastrectomy for cT3/4a Gastric Cancer (KLASS-10)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2023-0385
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Random group assignment during operation
  * Control group : Total omentectomy
  * Experimental group : Partial omentectomy Other surgical procedures are the same as usual in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total omentectomy group (Active Comparator): During minimally invasive radical gastrectomy and D2 lymph node dissection, total omentectomy will be performed.
  Interventions: Procedure: Arm I (Total omentectomy),
- Partial omentectomy group (Experimental): During minimally invasive radical gastrectomy and D2 lymph node dissection, partial omentectomy will be performed.
  Interventions: Procedure: Arm II (Partial omentectomy)

INTERVENTIONS:
Procedure: Arm I (Total omentectomy), — The surgery is performed with minimal invasive surgery, and the range of the surgery is radical gastrectomy and D2 lymph node dissection. Depending on the random assignment, total omentectomy and partial omentectomy (omentum preservation) will be performed for the control group and the experimental group, respectively. Total omentectomy removes whole greater omentum, while partial omentectomy preserves the omentum more than 3cm away from the gastro-epiploic vessels. Other surgical procedures are the same as usual in both groups.
  Arms: Total omentectomy group
Procedure: Arm II (Partial omentectomy) — The surgery is performed with minimal invasive surgery, and the range of the surgery is radical gastrectomy and D2 lymph node dissection. Depending on the random assignment, total omentectomy and partial omentectomy (omentum preservation) will be performed for the control group and the experimental group, respectively. Total omentectomy removes whole greater omentum, while partial omentectomy preserves the omentum more than 3cm away from the gastro-epiploic vessels. Other surgical procedures are the same as usual in both groups.
  Arms: Partial omentectomy group

SUMMARY:
For advanced gastric cancer, surgical resection is the only curable therapeutic strategy. According to minimally invasive approach is adopted in various field of oncologic surgery, laparoscopic gastrectomy with lymph node dissection is becoming a standard not only for early gastric cancer but also for advanced gastric cancer.

The greater omentum is an organ is known to play a role in removing bacteria in the abdominal cavity as a primary defense. Complete resection of the greater omentum has been considered essential to ensure the elimination of micrometastasis during surgery for advanced gastric cancer. However, the oncological effect of total omentectomy is still lack of evidence. Especially in minimal invasive gastrectomy, total omentectomy procedure is known to increases the operating time, increase the risk of bleeding, colonic injury, and postoperative complications such as intra-abdominal abscess, ascites, anastomotic leakage, ileus and wound infections. Therefore, in the case of minimal invasive surgery in early gastric cancer, omentectomy is omitted usually or routinely. Partial omentectomy preserves the omentum more than 3cm away from the gastro-epiploic vessels. Advanced energy devices facilitate partial omentectomy during laparoscopic gastrectomy.

According to the Japanese Gastric Cancer Treatment Guidelines, partial omentectomy (omentum preservation) is feasible for T1 or T2 tumors, and total omentectomy is recommended for clinical T3 or deeper tumors. However, the National Comprehensive Cancer Network(NCCN) guideline suggests total omentectomy and the European Society for Medical Oncology(ESMO) guideline does not mentioned about it.

It is still controversial whether total omentectomy should be performed in advanced gastric cancer. Therefore, we aimed to verify the non-inferiority of partial omentectomy, oncologic safety compared with total omentectomy via multicenter randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach
* Age between 20 to 85 years old
* ECOG PS 0-1, ASA class I-III
* Endoscopically Borrmann type I, II, III
* Clinical T3 and T4a tumors with or without regional lymph node metastases (cT3N0M0~T4aN3M0)
* Capable of minimal invasive radical subtotal gastrectomy with R0 resection in preoperative examinations
* Patients who signed an written consent form approved by the Institutional Review Board(IRB) after receiving sufficient explanations of the contents of the clinical trial
* Domestic patients who are able to follow up for 3 years after surgery

Exclusion Criteria:

* Confirmed distant metastasis in preoperative examinations
* Confirmed metastasis in abdominal cavity or distant organs during surgery
* Confirmed no infiltration of the serosa layer or unable to confirm the tumor location during surgery (sT1-2)
* Confirmed invasion of surrounding organs (sT4b)
* History of previous gastrectomy or greater omentum related surgery
* Patients who underwent preoperative treatment (chemotherapy, radiotherapy, or endoscopic submucosal dissection) for recently diagnosed gastric cancer
* Synchronous or metachronous malignancies, which underwent surgery, chemotherapy or radiotherapy within 5 years
* Patients judged to be inappropriate for the study by the physician. (ex. Pregnancy)
* Patients refused to participate after random assignment
* Surgery is not performed until 30 days after consenting to participate
* Patients who has participated in another on-going clinical trial, which is related surgical procedures and survival.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
3-year relapse free survival | 3 year after surgery
  Verify the non-inferiority of partial omentectomy(omentum preservation) in 3-year relapse free survival(RFS). Kaplan-Meier and log-rank tests will be used.

SECONDARY OUTCOMES:
3-year overall survival | 3 year after surgery
  To compare surgical outcomes between the partial omentectomy and total omentectomy in patients with advanced gastric cancer, especially clinical T3 and T4a tumors without distant metastasis, who underwent minimal invasive radical gastrectomy and D2 lymph node dissection.
  Clinicopathologic features and surgical outcomes will be analyzed using an paired t-test for continuous variables and the Chi-square test or Fisher's exact test for nominal variables. In the survival analysis, the Kaplan-Meier and log-rank tests will be used. Surgical complications will be graded according to the Clavien-Dindo classification.
Estimated blood loss | during surgery
  To compare surgical outcomes between the partial omentectomy and total omentectomy in patients with advanced gastric cancer, especially clinical T3 and T4a tumors without distant metastasis, who underwent minimal invasive radical gastrectomy and D2 lymph node dissection.
  Clinicopathologic features and surgical outcomes will be analyzed using an paired t-test for continuous variables and the Chi-square test or Fisher's exact test for nominal variables. In the survival analysis, the Kaplan-Meier and log-rank tests will be used. Surgical complications will be graded according to the Clavien-Dindo classification.
Operation time | during surgery
  To compare surgical outcomes between the partial omentectomy and total omentectomy in patients with advanced gastric cancer, especially clinical T3 and T4a tumors without distant metastasis, who underwent minimal invasive radical gastrectomy and D2 lymph node dissection.
  Clinicopathologic features and surgical outcomes will be analyzed using an paired t-test for continuous variables and the Chi-square test or Fisher's exact test for nominal variables. In the survival analysis, the Kaplan-Meier and log-rank tests will be used. Surgical complications will be graded according to the Clavien-Dindo classification.
Post-operative complications (Early, and delayed complication) | 1 month after surgery & 3 year after surgery ( Evaluate 2 times to analyze early complication, and delayed complication respectively)
  To compare surgical outcomes between the partial omentectomy and total omentectomy in patients with advanced gastric cancer, especially clinical T3 and T4a tumors without distant metastasis, who underwent minimal invasive radical gastrectomy and D2 lymph node dissection.
  Clinicopathologic features and surgical outcomes will be analyzed using an paired t-test for continuous variables and the Chi-square test or Fisher's exact test for nominal variables. In the survival analysis, the Kaplan-Meier and log-rank tests will be used. Surgical complications will be graded according to the Clavien-Dindo classification.
Post-operative mortality | 3 months after surgery
  To compare surgical outcomes between the partial omentectomy and total omentectomy in patients with advanced gastric cancer, especially clinical T3 and T4a tumors without distant metastasis, who underwent minimal invasive radical gastrectomy and D2 lymph node dissection.
  Clinicopathologic features and surgical outcomes will be analyzed using an paired t-test for continuous variables and the Chi-square test or Fisher's exact test for nominal variables. In the survival analysis, the Kaplan-Meier and log-rank tests will be used. Surgical complications will be graded according to the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No